CLINICAL TRIAL: NCT06345456
Title: Assessment of End-Tidal CO2 Levels in Patients Presenting to the Emergency Department With Gastrointestinal Bleeding
Brief Title: The Value of End-tidal Capnography in Gastrointestinal Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Emine Kilinc, medicine doctor, Izmir Katip Celebi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: izmirkatip
Record Dates: First submitted 2024-02-22; First posted 2024-04-03 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Gastro Intestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capnography device (Experimental)
  Interventions: Device: End-tidal capnography

INTERVENTIONS:
Device: End-tidal capnography — The value of end-tidal capnography

SUMMARY:
Gastrointestinal bleeding is a condition that frequently presents to emergency departments and can be fatal if diagnosis and treatment are delayed. The working mechanism of end tidal capnography is simply to detect the respiratory carbon dioxide level.

In our study, the investigators aimed to determine the severity of gastrointestinal bleeding by using the Glaskow Blachford Score and AIMS65 score in cases presenting with gastrointestinal bleeding, to determine the end tidal carbon dioxide value by capnography in these cases and to determine its effectiveness in evaluating mortality and morbidity in gastrointestinal bleeding.

DETAILED DESCRIPTION:
Gastrointestinal (GI) bleeding is a condition that frequently presents to emergency departments and has a mortal course in case of delayed diagnosis and treatment. Upper GI bleeding accounts for 5% of emergency department admissions. Mortality rates vary between 2% and 15%. Mostly, GI bleeding stops spontaneously and does not require endoscopic intervention, blood transfusion or surgery. However, among patients with life-threatening bleeding, timely intervention is very important. For this purpose, there are widely used and validated risk stratification tools such as the Glasgow Blatchford Score (GBS) and the AIMS65 score.

Capnography involves the noninvasive measurement of CO2 partial pressure during the respiratory cycle. It provides information on ventilation (efficiency of carbon dioxide elimination), perfusion (vascular CO2 transport) and metabolism (CO2 production through cellular metabolism). The principle of end-tidal capnography (ETCO2) is to detect the level of carbon dioxide in the expiratory breath.ETCO2 waveform changes provide information to physicians in various situations such as assessment of disease severity, cardiac arrest (quality of compression, return of spontaneous circulation, endotracheal tube placement, prognosis) procedural sedation and prediction of critical illness.

In our study, the investigators aimed to determine the relationship of ETCO2 value with GBS and AIMS65 scores and its effectiveness on the evaluation of morbidity and mortality in patients admitted to the emergency department with GI bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency department with symptoms and signs of gastrointestinal bleeding (hematochezia, melena, hematemesis).
* Patients with a presumptive diagnosis of gastrointestinal bleeding confirmed by endoscopy and colonoscopy.
* Patients who consent to participate in the study.
* Patients aged 18 and older.

Exclusion Criteria:

* Patients without symptoms and signs of gastrointestinal bleeding.
* Patients with a presumptive diagnosis of gastrointestinal bleeding ruled out by endoscopy and colonoscopy.
* Patients with respiratory pathologies that increase CO2 levels (such as asthma, COPD, pneumonia, etc.).
* Patients referred from external centers and underwent ERT replacement.
* Patients with heart failure.
* Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
The correlation between ETCO2 value and mortality in patients with gastrointestinal bleeding will be investigated. | six months
  The correlation between ETCO2 value and mortality in patients with gastrointestinal bleeding will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Katip Çelebi Üniversitesi, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Hearnshaw SA, Logan RF, Lowe D, Travis SP, Murphy MF, Palmer KR. Acute upper gastrointestinal bleeding in the UK: patient characteristics, diagnoses and outcomes in the 2007 UK audit. Gut. 2011 Oct;60(10):1327-35. doi: 10.1136/gut.2010.228437. Epub 2011 Apr 13. PMID 21490373
- [Background] van Leerdam ME, Vreeburg EM, Rauws EA, Geraedts AA, Tijssen JG, Reitsma JB, Tytgat GN. Acute upper GI bleeding: did anything change? Time trend analysis of incidence and outcome of acute upper GI bleeding between 1993/1994 and 2000. Am J Gastroenterol. 2003 Jul;98(7):1494-9. doi: 10.1111/j.1572-0241.2003.07517.x. PMID 12873568
- [Background] Sugawa C, Steffes CP, Nakamura R, Sferra JJ, Sferra CS, Sugimura Y, Fromm D. Upper GI bleeding in an urban hospital. Etiology, recurrence, and prognosis. Ann Surg. 1990 Oct;212(4):521-6; discussion 526-7. doi: 10.1097/00000658-199010000-00014. PMID 2222017
- [Background] Chen IC, Hung MS, Chiu TF, Chen JC, Hsiao CT. Risk scoring systems to predict need for clinical intervention for patients with nonvariceal upper gastrointestinal tract bleeding. Am J Emerg Med. 2007 Sep;25(7):774-9. doi: 10.1016/j.ajem.2006.12.024. PMID 17870480
- [Background] Pang SH, Ching JY, Lau JY, Sung JJ, Graham DY, Chan FK. Comparing the Blatchford and pre-endoscopic Rockall score in predicting the need for endoscopic therapy in patients with upper GI hemorrhage. Gastrointest Endosc. 2010 Jun;71(7):1134-40. doi: 10.1016/j.gie.2010.01.028. PMID 20598244
- [Background] Dicu D, Pop F, Ionescu D, Dicu T. Comparison of risk scoring systems in predicting clinical outcome at upper gastrointestinal bleeding patients in an emergency unit. Am J Emerg Med. 2013 Jan;31(1):94-9. doi: 10.1016/j.ajem.2012.06.009. Epub 2012 Sep 20. PMID 23000328
- [Background] Yang HM, Jeon SW, Jung JT, Lee DW, Ha CY, Park KS, Lee SH, Yang CH, Park JH, Park YS; Daegu-Gyeongbuk Gastrointestinal Study Group (DGSG). Comparison of scoring systems for nonvariceal upper gastrointestinal bleeding: a multicenter prospective cohort study. J Gastroenterol Hepatol. 2016 Jan;31(1):119-25. doi: 10.1111/jgh.13057. PMID 26211939
- [Background] Saltzman JR, Tabak YP, Hyett BH, Sun X, Travis AC, Johannes RS. A simple risk score accurately predicts in-hospital mortality, length of stay, and cost in acute upper GI bleeding. Gastrointest Endosc. 2011 Dec;74(6):1215-24. doi: 10.1016/j.gie.2011.06.024. Epub 2011 Sep 10. PMID 21907980
- [Background] Hyett BH, Abougergi MS, Charpentier JP, Kumar NL, Brozovic S, Claggett BL, Travis AC, Saltzman JR. The AIMS65 score compared with the Glasgow-Blatchford score in predicting outcomes in upper GI bleeding. Gastrointest Endosc. 2013 Apr;77(4):551-7. doi: 10.1016/j.gie.2012.11.022. Epub 2013 Jan 26. PMID 23357496
- [Background] Tang Y, Shen J, Zhang F, Zhou X, Tang Z, You T. Scoring systems used to predict mortality in patients with acute upper gastrointestinal bleeding in the ED. Am J Emerg Med. 2018 Jan;36(1):27-32. doi: 10.1016/j.ajem.2017.06.053. Epub 2017 Jun 27. PMID 28673695
- [Background] Whitaker DK. Time for capnography - everywhere. Anaesthesia. 2011 Jul;66(7):544-9. doi: 10.1111/j.1365-2044.2011.06793.x. Epub 2011 May 31. No abstract available. PMID 21627625
- [Background] Kodali BS. Capnography outside the operating rooms. Anesthesiology. 2013 Jan;118(1):192-201. doi: 10.1097/ALN.0b013e318278c8b6. No abstract available. PMID 23221867
- [Background] Nassar BS, Schmidt GA. Capnography During Critical Illness. Chest. 2016 Feb;149(2):576-585. doi: 10.1378/chest.15-1369. Epub 2016 Jan 12. PMID 26447854

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT06345456/SAP_000.pdf
  • Informed Consent Form (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT06345456/ICF_001.pdf